CLINICAL TRIAL: NCT03015493
Title: Cervical Traction Combined With Neural Mobilization for Patients With Cervical Radiculopathy: A Randomized Controlled Trial.
Brief Title: Effectiveness of Cervical Traction and Neural Mobilization in Patients With Cervical Radiculopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Christos Savva (Other)
Responsible Party: Sponsor-Investigator, Christos Savva, Lecturer, European University Cyprus
Organization: European University Cyprus (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHR7
Record Dates: First submitted 2017-01-06; First posted 2017-01-10 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Cervical Radiculopathy
Keywords: Neck pain; Neurodynamics; Spinal manipulative therapy
MeSH Terms: conditions — Radiculopathy; Neck Pain | interventions — Traction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Neural mobilization and traction (Experimental): Patients in this group are treated with neural mobilization techniques combined with cervical traction
  Interventions: Other: Neural mobilization combined with traction
- Traction group (Experimental): Patients in this group are treated with cervical traction
  Interventions: Other: Traction
- Control group (No Intervention): Patients in this group comprise the control group and are not treated with any intervention

INTERVENTIONS:
Other: Neural mobilization combined with traction — Neural mobilization techniques combined with cervical traction for the cervical nerve roots
  Arms: Neural mobilization and traction
Other: Traction — Traction techniques for the cervical spine
  Arms: Traction group

SUMMARY:
The purpose of the study is to examine the effects of cervical traction with or without the addition of neural mobilization, in patients with cervical radiculopathy

DETAILED DESCRIPTION:
Background:Cervical radiculopathy (CR) is a disorder of the peripheral nervous system where the resulted cervical nerve root (CNR) pathology produces a chronic pain and disability. Based on some epidemiological findings, CR is a common clinical diagnosis since its annual incidence has been estimated to be 83 cases per 100,000, with an increased prevalence noted in the fifth decade of life. In addition, C6 and C7 nerve roots are most commonly involved in this disorder, mainly due to the high range of motion occurring between cervical vertebrae C5-C6 and C6-C7.

CR is caused by a disc herniation, or a space-occupying lesion that can result in CNR inflammation, impingement, or both. In normal situations, CNRs ensure the normal function of sensation, movement and motor coordination of the upper limb. Therefore, the development of CR can produce sensory and motor deficits in the involved limb, including pins and needles, numbness and muscle weakness, along with a neuropathic pain described as a burning or shooting pain. These symptoms lead patients to exhibit severe functional limitations such as difficulties to work, to sleep or to participate in hobbies. Studies on this topic identified several socioeconomic and psychological deficits, from lost work and wages to prolonged pain and impaired social functioning, leading patients with CR to express symptoms of anxiety and depression.

Treatment of CR has been the subject of debate between physiotherapists and researchers. Several non-operative treatment approaches have been advocated to reduce CR pain and their analgesic effect has been recognized in a number of randomized clinical trials with these in turn being analyzed in few systematic reviews. Based on these studies, patients with CR can benefit from a multimodal treatment approach including the application of postural education, cervical traction and manual therapy techniques (mobilization, thrust manipulation etc.) applied to the cervical spine. However the small number of these studies as well as their poor methodological quality due to the short-term follow ups, lack of patient's homogeneity, randomization or control group etc., raise several questions about the validity of research findings and therefore much more studies are necessary. Among manual therapy techniques that have been recommended to improve the patient's pain and functional limitations, neural mobilization (NM) has been advocated as an effective treatment option. NM introduced as an intervention for pain relief more than 25 years ago are techniques that involve a specific sequence of joint movements to mobilize the involved peripheral nerve in order to facilitate the reduced nerve gliding and reduced the increased neural mechanosensitivity.

The application of NM is common but since now little research attention has been given to support its usage in patients with CR. Recently, a case study and a randomized controlled study concluded that neural mobilization applied simultaneously with cervical traction can produce clinically meaningful improvements over a 4-week period, in terms of pain, disability, function, grip strength and cervical spine range of motion. However, both methodological designs did not allow determining whether NM provided these benefits. Thus, the purpose of the present study was to examine the effects of cervical traction with or without the addition of NM, in patients with CR.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral sensory and motor deficits including sharp pain, muscle weakness and numbness in the upper arm
* A positive result in a minimum three of four tests (Spurling's test, Distraction test, Upper Limb Neurodynamic Test 1 and ipsilateral cervical rotation of less than 60) of a clinical prediction rule. This clinical prediction rule has demonstrated 94% specificity (95% = 0.88 to 1.00), 24% sensitivity (95% = 0.05 to 0.43) and a positive likelihood ratio of 6.1 (95% = 2.0 to 18.6) when 3 of 4 items were positive

Exclusion Criteria:

* A current history of cervical myelopathy or signs of upper motor neuron disease
* Bilateral CR or other musculoskeletal conditions in the affected limb.
* Receive of any prescription or over-the-counter analgesia or anti-inflammatory medication during the prior two weeks

Ages: 22 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index | Change from baseline after 4 weeks

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | Change from baseline after 4 weeks
Patient-Specific Functional Scale | Change from baseline after 4 weeks
Grip strength measurement using a dynamometer | Change from baseline after 4 weeks
Measurement of cervical spine active range of motion using a universal goniometer | Change from baseline after 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chritos Savva, PhD, Principal Investigator — European University Cyprus

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Result] Young IA, Michener LA, Cleland JA, Aguilera AJ, Snyder AR. Manual therapy, exercise, and traction for patients with cervical radiculopathy: a randomized clinical trial. Phys Ther. 2009 Jul;89(7):632-42. doi: 10.2522/ptj.20080283. Epub 2009 May 21. PMID 19465371